CLINICAL TRIAL: NCT05563246
Title: KRAKEN: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Oral Once-Daily LY3473329 in Adults With Elevated Lipoprotein(a) at High Risk for Cardiovascular Events
Brief Title: A Study of LY3473329 in Adult Participants With Elevated Lipoprotein(a) at High Risk for Cardiovascular Events
Acronym: KRAKEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18495; J2O-MC-EKBC (Other: Eli Lilly and Company); 2022-501466-21-00 (EU CTIS Number)
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Lipoprotein Disorder
Keywords: Atherosclerotic cardiovascular disease; ASCVD; Dyslipidemia; Lipoprotein(a); Lp(a); Cardiovascular; Cardiovascular disease; Cholesterol; Hyperlipidemia
MeSH Terms: conditions — Atherosclerosis; Dyslipidemias; Cardiovascular Diseases; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10 mg LY3473329 (Experimental): Participants received 10 milligrams (mg) of LY3473329 administered orally once daily (QD) over a 12-week treatment period.
  Interventions: Drug: LY3473329
- 60 mg LY3473329 (Experimental): Participants received 60 mg of LY3473329 administered orally QD over a 12-week treatment period.
  Interventions: Drug: LY3473329
- 240 mg LY3473329 (Experimental): Participants received 240 mg of LY3473329 administered orally QD over a 12-week treatment period.
  Interventions: Drug: LY3473329
- Placebo (Placebo Comparator): Participants received a matching dose of placebo administered orally QD over a 12-week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3473329 — Administered orally
  Arms: 10 mg LY3473329; 240 mg LY3473329; 60 mg LY3473329
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of LY3473329 in adult participants with elevated Lp(a) at high risk for cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 40 years old
* Participants with Lp(a) ≥175 nmol/L at randomization, measured at the central laboratory.
* High risk for cardiovascular events defined as documented coronary artery disease (CAD), stroke, or peripheral artery disease or atherosclerotic cardiovascular disease (ASCVD) risk equivalents (familial hypercholesterolemia or type 2 diabetes).
* Participants on the following medications according to local practice must be on a stable regimen for at least 4 weeks prior to randomization and expected to remain on a stable regimen through the end of the post-treatment follow-up period.

  * lipid-lowering drugs
  * testosterone, estrogens, anti-estrogens, progestins, selective estrogen receptor modulators, or growth hormone
* Have a body mass index within the range 18.5 to 40 kilogram/square meter (kg/m²), inclusive.
* Males who agree to use highly effective or effective methods of contraception may participate in this trial.
* Women of childbearing potential (WOCBP) who agree to use highly effective or effective methods of contraception and women not of childbearing potential (WNOCBP) may participate in this trial.

Exclusion Criteria:

* Have a history or presence of an underlying disease, or surgical, physical, medical, or psychiatric condition that, in the opinion of the investigator, would potentially affect participant safety within the study or interfere with participating in or completing the study or with the interpretation of data.
* Any of the following, or other events indicating unstable medical condition in the opinion of the investigator, within 3 months of randomization:

  * major surgery
  * coronary, carotid, or peripheral arterial revascularization
  * stroke or transient ischemic attack
  * myocardial infarction or unstable angina
  * acute limb ischemia
* Have, in the 6 months prior to day 1, uncontrolled Type 1 or Type 2 diabetes
* Have uncontrolled hypertension

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (42):
- United States (3):
  - Care Access - Baltimore, Baltimore, Maryland
  - Care Access - Dorchester, Dorchester, Massachusetts
  - Care Access - Lima, Lima, Ohio
- Australia (4):
  - Core Research Group, Brisbane, Queensland
  - Nightingale Research, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Victorian Heart Hospital, Clayton, Victoria
- Brazil (8):
  - CEDOES, Vitória, Espírito Santo
  - Pesquisa Clínica em Diabetes - Dra Rosângela Réa, Curitiba, Paraná
  - Centro de Pesquisa Clinica do Coracao, Acaraju, Sergipe
  - Incor - Instituto do Coracao, São Paulo, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - CPCLIN, São Paulo
  - Instituto Dante Pazzanese de Cardiology, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- China (8):
  - Third People's Hospital of Hainan Province, Sanya, Hainan
  - The First Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Changzhou Second People's Hospital, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - China-Japan Union Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
- Germany (4):
  - Gemeinschaftpraxis Dr. med. Martin Prohaska und Dr. med. Felix Schulte, Mühldorf, Bavaria
  - ClinPhenomics GmbH & Co KG, Frankfurt am Main, Hesse
  - Kath. St.-Johannes-Gesellschaft Dortmund, Dortmund, North Rhine-Westphalia
  - Private Practice - Dr. Frank Menzel, Dessau
- Hungary (6):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged, Csongrád megye
  - Medifarma 98 Kft, Nyíregyháza, Nyíregyháza
  - Flor Ferenc Hospital of Pest County, Kistarcsa, Pest County
  - Belvárosi Egészségház, Zalaegerszeg, Zala County
  - Dél-Pesti Centrumkórház, Budapest
  - Semmelweis University, Budapest
- Japan (7):
  - Funabashi Municipal Medical Center, Funabashi, Chiba
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Minamino Cardiovascular Hospital, Hachiōji, Tokyo
  - Hiroshima City Hospital, Hiroshima
  - Miyazaki Medical Association Hospital, Miyazaki
- Netherlands (2):
  - VieCuri Medisch Centrum, locatie Venlo, Venlo, Limburg
  - Meander Medisch Centrum, Amersfoort, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Nicholls SJ, Ni W, Rhodes GM, Nissen SE, Navar AM, Michael LF, Haupt A, Krege JH. Oral Muvalaplin for Lowering of Lipoprotein(a): A Randomized Clinical Trial. JAMA. 2025 Jan 21;333(3):222-231. doi: 10.1001/jama.2024.24017. PMID 39556768
- [Derived] Nicholls SJ, Nelson AJ, Michael LF. Oral agents for lowering lipoprotein(a). Curr Opin Lipidol. 2024 Dec 1;35(6):275-280. doi: 10.1097/MOL.0000000000000953. Epub 2024 Sep 25. PMID 39329200
- [Derived] Karp A, Jacobs M, Barris B, Labkowsky A, Frishman WH. Lipoprotein(a): A Review of Risk Factors, Measurements, and Novel Treatment Modalities. Cardiol Rev. 2025 Jul-Aug 01;33(4):352-358. doi: 10.1097/CRD.0000000000000667. Epub 2024 Feb 28. PMID 38415744
- See also: A Study of LY3473329 in Adult Participants With Elevated Lipoprotein(a) at High Risk for Cardiovascular Events (KRAKEN) — https://trials.lilly.com/en-US/trial/362835

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 10 mg LY3473329 | 60 mg LY3473329 | 240 mg LY3473329 | Placebo
Started | 34 | 64 | 68 | 67
Received at Least One Dose of Study Drug | 34 | 63 | 68 | 67
Completed | 33 | 60 | 65 | 67
Not Completed | 1 | 4 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 10 mg LY3473329: Participants received 10 mg of LY3473329 administered orally QD over a 12-week treatment period.
- Total: Total of all reporting groups
Arm/Group | 10 mg LY3473329 | 60 mg LY3473329 | 240 mg LY3473329 | Placebo | Total
Number analyzed (Participants) | 34 | 64 | 68 | 67 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.06 (10.01) | 65.50 (9.36) | 64.75 (9.35) | 62.78 (9.93) | 64.29 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 22 | 24 | 19 | 76
  Male | 23 | 42 | 44 | 48 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 11 | 10 | 9 | 34
  Not Hispanic or Latino | 30 | 50 | 57 | 58 | 195
  Unknown or Not Reported | 0 | 3 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 17 | 19 | 18 | 63
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 2 | 5 | 1 | 1 | 9
  White | 22 | 41 | 45 | 45 | 153
  More than one race | 0 | 1 | 3 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 6 | 12 | 12 | 12 | 42
  Brazil | 6 | 13 | 12 | 12 | 43
  China | 4 | 8 | 9 | 9 | 30
  Germany | 4 | 5 | 8 | 7 | 24
  Hungary | 6 | 11 | 11 | 11 | 39
  Japan | 4 | 8 | 8 | 9 | 29
  Netherlands | 2 | 3 | 3 | 4 | 12
  United States | 2 | 4 | 5 | 3 | 14
Lp(a) - Assessed via Intact Lp(a) Assay [Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)] — Lipoprotein(a) [Lp(a)] levels were assessed using an assay that measured intact Lp(a) particles, referred to as the "intact Lp(a) assay." Population: All randomized participants who had non-missing baseline Lp(a) data, as assessed by the intact Lp(a) assay. As pre-specified in the statistical analysis plan, intact Lp(a) assay measurements were not collected from participants at Chinese sites due to country-specific restrictions on sample storage.
  nanomoles per liter (nmol/L)
    number analyzed (Participants) | 28 | 52 | 57 | 57 | 194
    (all) | 220.99 (60.39) | 223.47 (97.36) | 242.42 (100.18) | 250.53 (96.66) | 236.63 (93.74)
Lp(a) - Assessed via Apo(a) Assay [Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)] — Lp(a) levels were assessed using an assay that measured total apolipoprotein(a) [apo(a)], referred to as the "apo(a) assay." Population: All randomized participants who had non-missing baseline Lp(a) data, as assessed by the apo(a) assay.
  nanomoles per liter (nmol/L)
    number analyzed (Participants) | 34 | 63 | 68 | 67 | 232
    (all) | 269.67 (78.10) | 256.28 (96.55) | 273.84 (90.68) | 265.30 (85.80) | 265.99 (88.93)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lp(a) - Assessed Via Intact Lp(a) Assay
Description: Least Squares Mean (LS Mean) was calculated using a Mixed Model for Repeated Measures (MMRM): Log (Actual Measurement/Baseline) = Log (Baseline) + Country + Treatment + Time + Treatment*Time.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug had a non-missing baseline value and at least one post-baseline value, as assessed by the intact Lp(a) assay, excluding data after discontinuation of the study drug or initiation of new Lp(a) modifying medication. As pre-specified in the statistical analysis plan, intact Lp(a) assay measurements were not collected from participants at Chinese sites due to country-specific restrictions on sample storage.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 10 mg LY3473329 | 60 mg LY3473329 | 240 mg LY3473329 | Placebo
Number analyzed (Participants) | 23 | 45 | 47 | 49
Percent change | -47.35 (4.811) | -81.57 (1.230) | -85.71 (0.927) | 0.48 (6.382)
Statistical Analysis 1: Comparison: 10 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference (Final Values) = -47.61, 95% CI 2-sided [-57.68 to -35.14]
Statistical Analysis 2: Comparison: 60 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference (Final Values) = -81.66, 95% CI 2-sided [-84.62 to -78.13]
Statistical Analysis 3: Comparison: 240 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference (Final Values) = -85.77, 95% CI 2-sided [-88.03 to -83.09]

2. Primary Outcome: Percent Change From Baseline in Lp(a) - Assessed Via Apo(a) Assay
Description: LS Mean was calculated using a MMRM: Log (Actual Measurement/Baseline) = Log (Baseline) + Country + Treatment + Time + Treatment*Time.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug, had a non-missing baseline value, and at least one post-baseline value, as assessed by the apo(a) assay, excluding data after discontinuation of the study drug or initiation of new Lp(a) modifying medication.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 10 mg LY3473329 | 60 mg LY3473329 | 240 mg LY3473329 | Placebo
Number analyzed (Participants) | 29 | 56 | 57 | 60
Percent change | -42.26 (4.477) | -70.90 (1.669) | -69.88 (1.676) | -3.15 (5.342)
Statistical Analysis 1: Comparison: 10 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference (Final Values) = -40.38, 95% CI 2-sided [-50.45 to -28.27]
Statistical Analysis 2: Comparison: 60 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference (Final Values) = -69.95, 95% CI 2-sided [-74.23 to -64.96]
Statistical Analysis 3: Comparison: 240 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference (Final Values) = -68.90, 95% CI 2-sided [-73.27 to -63.81]

3. Secondary Outcome: Percentage of Participants Who Achieved Lp(a) < 125 Nmol/L - Assessed Via Intact Lp(a) Assay
Description: The percentage of participants who achieved Lp(a) less than (<) 125 nmol/L, as measured using the intact Lp(a) assay, with data analysis performed through a logistic regression model that included imputed missing values, was reported.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of the study drug and had a non-missing baseline value, as assessed by the intact Lp(a) assay, excluding data after discontinuation of the study drug or initiation of new Lp(a) modifying medication. As pre-specified in the statistical analysis plan, intact Lp(a) assay measurements were not collected from participants at Chinese sites due to country-specific restrictions on sample storage.
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg LY3473329 | 60 mg LY3473329 | 240 mg LY3473329 | Placebo
Number analyzed (Participants) | 23 | 45 | 47 | 49
Percentage of participants | 69.6 | 95.6 | 95.7 | 6.1
Statistical Analysis 1: Comparison: 10 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Regression, Logistic; Risk Difference (RD) = 58.15, 95% CI 2-sided [40.30 to 75.99]
Statistical Analysis 2: Comparison: 60 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Regression, Logistic; Risk Difference (RD) = 89.87, 95% CI 2-sided [81.54 to 98.20]
Statistical Analysis 3: Comparison: 240 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Regression, Logistic; Risk Difference (RD) = 90.71, 95% CI 2-sided [82.80 to 98.62]

4. Secondary Outcome: Percentage of Participants Who Achieved Lp(a) < 125 Nmol/L - Assessed Via Apo(a) Assay
Description: The percentage of participants who achieved Lp(a) < 125 nmol/L, as measured using the apo(a) assay, with data analysis performed through a logistic regression model that included imputed missing values, was reported.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of the study drug and had a non-missing baseline value, as assessed by the apo(a) assay, excluding data after discontinuation of the study drug or initiation of new Lp(a) modifying medication.
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg LY3473329 | 60 mg LY3473329 | 240 mg LY3473329 | Placebo
Number analyzed (Participants) | 29 | 56 | 57 | 60
Percentage of participants | 37.9 | 82.1 | 77.2 | 3.3
Statistical Analysis 1: Comparison: 10 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Regression, Logistic; Risk Difference (RD) = 35.18, 95% CI 2-sided [18.90 to 51.46]
Statistical Analysis 2: Comparison: 60 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Regression, Logistic; Risk Difference (RD) = 78.18, 95% CI 2-sided [67.70 to 88.65]
Statistical Analysis 3: Comparison: 240 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Regression, Logistic; Risk Difference (RD) = 73.62, 95% CI 2-sided [63.65 to 83.58]

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB)
Description: LS Mean was calculated using a MMRM: Log (Actual Measurement/Baseline) = Log (Baseline) + Country + Baseline Lp(a) Stratum + Treatment + Time + Treatment*Time.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug and had a non-missing baseline value and at least one post-baseline value for this outcome, excluding data after discontinuation of the study drug or initiation of new Lp(a) modifying medication.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 10 mg LY3473329 | 60 mg LY3473329 | 240 mg LY3473329 | Placebo
Number analyzed (Participants) | 29 | 56 | 57 | 60
Percent change | -10.49 (4.349) | -14.53 (3.055) | -17.56 (2.877) | -1.70 (3.362)
Statistical Analysis 1: Comparison: 10 mg LY3473329 vs Placebo; Test type: Superiority; p = 0.110, Mixed Models Analysis; LS Mean Difference (Final Values) = -8.94, 95% CI 2-sided [-18.84 to 2.17]
Statistical Analysis 2: Comparison: 60 mg LY3473329 vs Placebo; Test type: Superiority; p = 0.004, Mixed Models Analysis; LS Mean Difference (Final Values) = -13.05, 95% CI 2-sided [-20.92 to -4.40]
Statistical Analysis 3: Comparison: 240 mg LY3473329 vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; LS Mean Difference (Final Values) = -16.13, 95% CI 2-sided [-23.69 to -7.84]

6. Secondary Outcome: Percent Change From Baseline in High-Sensitivity C-Reactive Protein (hsCRP)
Description: as for outcome 5
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 10 mg LY3473329 | 60 mg LY3473329 | 240 mg LY3473329 | Placebo
Number analyzed (Participants) | 29 | 56 | 57 | 58
Percent change | 21.87 (20.029) | -2.41 (11.713) | -15.39 (9.921) | -9.91 (10.526)
Statistical Analysis 1: Comparison: 10 mg LY3473329 vs Placebo; Test type: Superiority; p = 0.131, Mixed Models Analysis; LS Mean Difference (Final Values) = 35.27, 95% CI 2-sided [-8.63 to 100.27]
Statistical Analysis 2: Comparison: 60 mg LY3473329 vs Placebo; Test type: Superiority; p = 0.627, Mixed Models Analysis; LS Mean Difference (Final Values) = 8.32, 95% CI 2-sided [-21.62 to 49.70]
Statistical Analysis 3: Comparison: 240 mg LY3473329 vs Placebo; Test type: Superiority; p = 0.701, Mixed Models Analysis; LS Mean Difference (Final Values) = -6.08, 95% CI 2-sided [-31.89 to 29.51]

7. Secondary Outcome: Pharmacokinetics (PK): Trough Concentrations (C-trough) of LY3473329
Description: C-trough were measured at specified time points to assess the minimum concentration of LY3473329 in the blood before the next dose was administered.
Time Frame: Week from randomization 1, 2, 8, 12: Pre-dose
Population: All randomized participants who received at least one dose of the study drug and had evaluable PK samples for the relevant weeks were included in this outcome analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 10 mg LY3473329 | 60 mg LY3473329 | 240 mg LY3473329
Number analyzed (Participants) | 33 | 60 | 66
nanograms per milliliter (ng/mL)
  Week 1: number analyzed (Participants) | 33 | 59 | 64
  Week 1 | 13.0 (81) | 42.4 (79) | 83.3 (70)
  Week 2: number analyzed (Participants) | 31 | 59 | 66
  Week 2 | 14.8 (73) | 39.3 (76) | 77.9 (62)
  Week 8: number analyzed (Participants) | 32 | 59 | 62
  Week 8 | 14.5 (67) | 38.8 (89) | 73.9 (110)
  Week 12: number analyzed (Participants) | 31 | 60 | 63
  Week 12 | 15.4 (64) | 37.7 (95) | 74.0 (111)

ADVERSE EVENTS:
Time Frame: Baseline to end of follow-up (up to 16 weeks)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | 10 mg LY3473329 | 60 mg LY3473329 | 240 mg LY3473329 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/63 | 0/68 | 0/67
Serious Adverse Events (participants affected / at risk) | 2/34 | 2/63 | 2/68 | 4/67
Other Adverse Events (participants affected / at risk) | 7/34 | 5/63 | 10/68 | 11/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 10 mg LY3473329 (N=34) | 60 mg LY3473329 (N=63) | 240 mg LY3473329 (N=68) | Placebo (N=67)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0/23 (0) | 0/41 (0) | 1/44 (1) | 0/48 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 10 mg LY3473329 (N=34) | 60 mg LY3473329 (N=63) | 240 mg LY3473329 (N=68) | Placebo (N=67)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 4 (4) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/11 (0) | 0/22 (0) | 0/24 (0) | 1/19 (1)

LIMITATIONS AND CAVEATS:
Due to country-specific restrictions on sample storage, measurements for the primary endpoint and key secondary endpoints involving Lp(a), as assessed by the intact Lp(a) assay, could not be obtained from participants at the Chinese sites. As a result, intact Lp(a) assay outcome data from these sites were not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT05563246/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT05563246/SAP_001.pdf